CLINICAL TRIAL: NCT01575132
Title: STN-DBS Retrospective/Prospective Study With a Follow-up Time of Minimum 10 Years
Brief Title: Deep Brain Stimulation Follow-up After 10 Years
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-106-12
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Stimulation, Deep Brain; Study, Follow-Up; Adverse Effects
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's Disease, DBS, 10-14 years

SUMMARY:
The purpose of this study is to examine the long-term effect of Deep Brain Stimulation (DBS) for patients with Parkinson's Disease. We have data for patients operated with DBS since 1998. We wish to examine the effect of stimulation on motor symptoms as well as make a follow-up on complications and side-effects related to treatment. We also wish to follow-up on the quality of life-studies made in the years 2003-2008.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is caused by a progressive loss of dopamine-producing cells in substantia nigra in mesencephalon.

PD is characterized by the symptoms resting tremor, rigidity and bradykinesia. Later in the course of the disease, patients develop gait- and balance symptoms. In the first years of the disease, the patients' symptoms are treated well with levodopa. As the disease develops and the loss of dopamine-producing cells grows, the physiological buffer-capacity for levodopa is lost and patients develop motor fluctuations in the shape of on-off symptoms and dyskinesias. Patients with these symptoms may benefit from implantation of electrodes in the subthalamic nucleus, which is stimulated by an pulse generator on the chest.

A number of studies have found a long-term effect of DBS, but most of these studies have a follow-up time of no more than five years. Overall, these studies show a beneficial effect of DBS after five years: The patients need less medication, the number of off-periods is decreased and they score lower on the Unified Parkinson Disease Rating Scale, part three. However, the axial symptoms and the bradykinesia progress.

As of yet, few studies examine the effect of Deep Brain Stimulation after 10 years. In our study we wish to examine the effect of DBS for all patients operated at Aarhus University Hospital in the years 1998-2002, which gives us a follow-up time of 10-14 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease treated with DBS at Aarhus University Hospital in the years 1998-2002.

Exclusion Criteria:

* Dementia, i.e. MMSE<24
* DBS removed
* Deceased

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Parkinson-patients treated with Deep Brain Stimulation at Aarhus University Hospital in the years 1998-2002.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-04 (Estimated); Study Completion 2015-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ostergaard, DMSci, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Neurology, Aarhus, Denmark